CLINICAL TRIAL: NCT03777761
Title: A Phase 1, Randomized, Partially Double-Blind, Placebo- and Positive-controlled Study to Evaluate the Effect of Tucatinib on Cardiac Repolarization in Healthy Subjects
Brief Title: Effects of Tucatinib on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ONT-380-011
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — tucatinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be double-blind in regard to tucatinib and placebo study treatments and open-label for the positive control, moxifloxacin.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): tucatinib + placebo + moxifloxacin (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin
- Treatment Sequence CAB (Experimental): moxifloxacin + tucatinib + placebo (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin
- Treatment Sequence BCA (Experimental): placebo + moxifloxacin + tucatinib (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin
- Treatment Sequence CBA (Experimental): moxifloxacin + placebo + tucatinib (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin
- Treatment Sequence ACB (Experimental): tucatinib + moxifloxacin + placebo (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin
- Treatment Sequence BAC (Experimental): placebo + tucatinib + moxifloxacin (administered in sequential treatment periods)
  Interventions: Drug: tucatinib; Drug: placebo; Drug: moxifloxacin

INTERVENTIONS:
Drug: tucatinib — 300mg oral dose
Drug: placebo — Matching placebo for tucatinib
Drug: moxifloxacin — 400mg single oral dose

SUMMARY:
This study is looking at how the study drug, tucatinib, affects the heart. Tucatinib is being studied as a possible treatment for breast cancer. This study will recruit healthy volunteers. There are 3 parts in the study. Each volunteer will be in all 3 parts. One part will be to take the study drug, the second part will be to take a placebo (pill with no medicine), and the third part will be to take moxifloxacin. The volunteers will only know what part of the study they are in when they take moxifloxacin. For the study drug and placebo parts, volunteers will take 2 pills by mouth for 5 days. For the moxifloxacin part, volunteers will take 1 pill by mouth for 1 day.

DETAILED DESCRIPTION:
This study will evaluate the effects of a steady state therapeutic dose of tucatinib on QTcF (QT interval corrected for heart rate using Fridericia's method) in healthy individuals. In this design, study treatment will be dosed in 3 sequential treatment periods:

Treatment A: Oral doses of 300mg tucatinib for 5 days

Treatment B: Oral doses of matching placebo for tucatinib for 5 days

Treatment C: A single oral dose of 400 mg of moxifloxacin

Patients will be randomized based on 2-Williams-square design to 1 of 6 treatment sequences to maintain the study blind for tucatinib and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Good health, determined by medical history, physical examination, 12-lead ECG, vital signs measurements, or clinical laboratory evaluations
* Body mass index (BMI) between 18 and 32 kg/m^2
* Body weight between 50 and 100 kg
* Female subjects must be of non-childbearing potential
* Male subjects must agree to use contraception or be surgically sterile for at least 90 days

Exclusion Criteria:

* Significant history of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Any condition affecting drug absorption
* History of hypersensitivity or allergy to any drug compound, food, or other substance
* Single 12-lead ECG demonstrating QTcF >450 msec for males or >470 msec for females, or history/evidence of long QT syndrome
* History of alcoholism or drug/chemical abuse within 2 years
* Use of prescription products within 30 days prior to check in
* Use of nonprescription products within 14 days prior to check in, including vitamins, minerals, and herbal supplements
* Use of tobacco- or nicotine-containing products within 3 months prior to check in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change-from-baseline in QTcF | Up to 32 days
  QTcF is the QT interval corrected for heart rate using Fridericia's method.

SECONDARY OUTCOMES:
Change from baseline in heart rate (HR) | Up to 32 days
Change from baseline in QTcF | Up to 32 days
Change from baseline in PR interval | Up to 32 days
Change from baseline in QRS interval | Up to 32 days
Placebo-corrected change from baseline in HR | Up to 32 days
Placebo-corrected change from baseline in PR interval | Up to 32 days
Placebo-corrected change from baseline in QRS interval | Up to 32 days
• Number of participants who experience increases in absolute QTcF interval values >450 msec | Up to 32 days
• Number of participants who experience QTcF interval changes from predose baseline of >30msec | Up to 32 days
• Number of participants who experience an increase in PR interval from predose baseline of >25% to a PR >200 msec | Up to 32 days
• Number of participants who experience an increase in QRS interval from predose baseline >25% to a QRS >120 msec | Up to 32 days
• Number of participants who experience a decrease in heart rate >25% from baseline to a heart rate <50 | Up to 32 days
• Number of participants who experience an increase in heart rate >25% from baseline to a heart rate >100 | Up to 32 days
Frequency of treatment-emergent changes of T-wave morphology and U-wave presence | Up to 32 days
Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUC[0-inf]) for tucatinib and ONT-993 | Up to 26 days
AUC from time 0 to the time of the last quantifiable concentration for tucatinib and ONT-993 | Up to 26 days
Percentage of AUC[0-inf] due to extrapolation for tucatinib and ONT-993 | Up to 26 days
Maximum observed concentration for tucatinib and ONT-993 | Up to 26 days
Time of maximum observed concentration for tucatinib and ONT-993 | Up to 26 days
Apparent terminal elimination half-life for tucatinib and ONT-993 | Up to 26 days
Apparent total clearance for tucatinib | Up to 26 days
Apparent volume of distribution during the terminal phase for tucatinib | Up to 26 days
Metabolic ratio based on AUC for ONT-993 | Up to 26 days
Incidence of adverse events (AEs) | Up to 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Woolery, PharmD, BCOP, Study Director — Seagen Inc.
Locations (1):
- Covance Clinical Research Unit - Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Topletz-Erickson AR, Mayor JG, Liu HT, Abdulrasool LI, Endres CJ. Effect of Tucatinib on Cardiac Repolarization in Healthy Volunteers. Drugs R D. 2023 Dec;23(4):411-419. doi: 10.1007/s40268-023-00440-8. Epub 2023 Sep 26. PMID 37751113